CLINICAL TRIAL: NCT00262925
Title: A Phase II Study of MOAD (Methotrexate, Vincristine, L-asparaginase and Dexamethasone) With Subcutaneous Campath for Adults With Relapsed or Refractory Acute Leukemia (ALL)
Brief Title: Combination Chemotherapy and Alemtuzumab in Treating Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00518; E1904 (Other: Eastern Cooperative Oncology Group); U10CA021115 (NIH)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Adult Acute Lymphoblastic Leukemia
Keywords: MOAD; Methotrexate; Vincristine; L-asparaginase; Dexamethasone; Subcutaneous Campath
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Alemtuzumab; Asparaginase; palmitoyl-L-asparaginase; Methotrexate; merphos; Dexamethasone; Calcium Dobesilate; Leucovorin; Mercaptopurine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy, enzyme inhibitor therapy) (Experimental): INDUCTION THERAPY: Patients receive methotrexate IV; vincristine IV and asparaginase IM ; oral dexamethasone ; and alemtuzumab SC.
  CONSOLIDATION THERAPY: Patients receive methotrexate IV and asparaginase IM.
  CYTOREDUCTION THERAPY: Patients receive vincristine IV and methotrexate IV; leucovorin calcium IV; and oral dexamethasone.
  MAINTENANCE THERAPY: Patients receive oral mercaptopurine; oral methotrexate; vincristine IV; and oral dexamethasone.
  Interventions: Biological: alemtuzumab; Drug: asparaginase; Drug: methotrexate; Drug: dexamethasone; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: vincristine

INTERVENTIONS:
Biological: alemtuzumab — Given subcutaneously
  Other Names: anti-CD52 monoclonal antibody; Campath-1H; MoAb CD52; Monoclonal Antibody Campath-1H; Monoclonal Antibody CD52
Drug: asparaginase — Given IM
  Other Names: ASNase; Colaspase; Crasnitin; Elspar; L-ASP
Drug: methotrexate — Given IV or orally
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: dexamethasone — Given orally
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: mercaptopurine — Given orally
  Other Names: 6-mercaptopurine; 6-MP; Leukerin; MP
Drug: vincristine — Given IV
  Other Names: vincristine sulfate; leurocristine sulfate; VCR; Vincasar PFS

SUMMARY:
This phase II trial is studying how well giving combination chemotherapy together with alemtuzumab works in treating patients with relapsed or refractory acute lymphoblastic leukemia. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Monoclonal antibodies, such as alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving combination chemotherapy together with alemtuzumab may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the complete response rate in patients with relapsed or refractory acute lymphoblastic leukemia treated with methotrexate, vincristine, asparaginase, and dexamethasone (MOAB) in combination with alemtuzumab.

II. Determine disease-free and/or overall survival of patients treated with this regimen.

III. Determine the toxic effects of this regimen in these patients.

IV. Correlate the density of cluster of differentiation 52 (CD52) molecules on the surface of leukemic lymphoblasts with response in patients treated with this regimen.

V. Correlate the presence of minimal residual disease at the time of maximal response to this regimen with overall outcome in these patients.

OUTLINE: This is a multicenter study. The study had two steps. Step 1: 5 mg dose of Campath (alemtuzumab); Step 2: 10 mg dose of Campath.

INDUCTION THERAPY: Patients receive methotrexate intravenously (IV) on day 1; vincristine IV and asparaginase intramuscularly (IM) on day 2; oral dexamethasone on days 1-10; and alemtuzumab subcutaneously (SC) on days 1, 4, and 7. Treatment repeats every 10 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete remission (CR) proceed to consolidation therapy.

CONSOLIDATION THERAPY: Patients receive methotrexate IV on day 1 and asparaginase IM on day 2. Treatment repeats every 10 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients who remain in CR proceed to cytoreduction therapy.

CYTOREDUCTION THERAPY: Patients receive vincristine IV and methotrexate IV over 6 hours on day 1; leucovorin calcium IV continuously over 24 hours on days 1 and 2 and then orally 4 times a day on day 3; and oral dexamethasone on days 2-6. Treatment repeats every 30 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients who remain in CR proceed to maintenance therapy.

MAINTENANCE THERAPY: Patients receive oral mercaptopurine on days 1-30; oral methotrexate on days 1, 8, 15, and 22; vincristine IV on day 1; and oral dexamethasone on days 1-5. Treatment repeats every 30 days for 36 courses in the absence of disease progression or unacceptable toxicity.

Patients are assessed every 3 months if patient is < 2 years from study entry and every 6 months if patient is 2-5 years from study entry.

PROJECTED ACCRUAL: Allowing for two dose levels, a maximum of 48 patients may be accrued approximately in 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or relapsed acute lymphoblastic leukemia

  * Must be in first relapse or have failed to achieve complete remission with 1 prior regimen
* Prior central nervous system (CNS) leukemia allowed provided cerebrospinal fluid is normal
* ECOG Performance status of 0-3
* Bilirubin normal
* Creatinine normal
* Human immunodeficiency virus (HIV) negative
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Hepatitis B positivity
* Bacterial or fungal infection
* Infection requiring treatment with antibiotics
* Active cytomegalovirus infection by molecular detection methods
* Known hypersensitivity to alemtuzumab or its components
* Pregnant or nursing
* Other malignancy within the past 5 years except adequately treated basal cell skin cancer or cervical carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-06; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wiernik, Principal Investigator — Montefiore Medical Center
Locations (58):
- United States (58):
  - Rush - Copley Medical Center, Aurora, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Saint Anthony Memorial Health Center, Michigan City, Indiana
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor Therapy)
Started | 12 (7 patients were enrolled to step 1, and 5 patients were enrolled to step 2)
Completed | 1
Not Completed | 11
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 4
Not completed — Death | 2
Not completed — alternative therapy | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients, and 7 were entered to the first step with 5mg Campath dose, 5 entered to the second step with 10mg Campath dose
Groups:
- Treatment (Chemotherapy, Enzyme Inhibitor Therapy): INDUCTION THERAPY: Patients receive methotrexate IV; vincristine IV and asparaginase IM; oral dexamethasone; and alemtuzumab SC on days 1, 4, and 7.
  CONSOLIDATION THERAPY: Patients receive methotrexate IV and asparaginase IM.
  CYTOREDUCTION THERAPY: Patients receive vincristine IV and oral methotrexate IV; leucovorin calcium IV; and oral dexamethasone.
  MAINTENANCE THERAPY: Patients receive oral mercaptopurine; oral methotrexate; vincristine IV; and oral dexamethasone.
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 12
Age, Customized [Median (Full Range); unit: years] | 35 [19 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Complete response requires that all of the following be present for at least four weeks.
  1. Peripheral Blood Counts: Neutrophil count >= 1.0 x 109/L, Platelet count >= 100 x 109/L, Reduced hemoglobin concentration or hematocrit has no bearing on remission status, Leukemic blasts must not be present in the peripheral blood.
  2 .Bone Marrow Aspirate and Biopsy: Cellularity of bone marrow biopsy must be > 20% with maturation of all cell lines, <= 5% blasts.
  3. Extramedullary leukemia, such as CNS or soft tissue involvement, must not be present.
Time Frame: assessed before the first consolidation cycle and first cytoreduction cycle, before the first and after the last maintenance cycle; after discontinuing treatment, assessed every 3 months if < 2 years and every 6 months if 2-5 years from study entry
Population: all enrolled patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 12
percentage of participants | 33 [10 to 65]

2. Secondary Outcome: Overall Survival
Description: Time from registration to death from any cause. Patients alive were censored at follow up.
Time Frame: assessed every 3 months if patient is < 2 years from study entry and every 6 months if patient is 2-5 years from study entry
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment (Chemotherapy, Enzyme Inhibitor Therapy): Detailed Description Section
  INDUCTION THERAPY: Patients receive methotrexate IV; vincristine IV and asparaginase IM; oral dexamethasone; and alemtuzumab SC on days 1, 4, and 7.
  CONSOLIDATION THERAPY: Patients receive methotrexate IV and asparaginase IM.
  CYTOREDUCTION THERAPY: Patients receive vincristine IV and oral methotrexate IV; leucovorin calcium IV; and oral dexamethasone.
  MAINTENANCE THERAPY: Patients receive oral mercaptopurine; oral methotrexate; vincristine IV; and oral dexamethasone.
  alemtuzumab: Given subcutaneously
  asparaginase: Given IM
  methotrexate: Given IV or orally
  dexamethasone: Given orally
  leucovorin calcium: Given IV
  mercaptopurine tablet: Given orally
  vincristine sulfate: Given IV
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 12
months | 5.2 [0.76 to 21]

ADVERSE EVENTS:
Time Frame: Assessed every while on treatment and for 30 days after the end of treatment
Groups:
- MOAD+Campath-Step 1: Campath 5mg dose
  INDUCTION THERAPY: Patients receive methotrexate IV; vincristine IV and asparaginase IM; oral dexamethasone; and alemtuzumab SC.
  CONSOLIDATION THERAPY: Patients receive methotrexate IV and asparaginase IM.
  CYTOREDUCTION THERAPY: Patients receive vincristine IV and oral methotrexate IV; leucovorin calcium IV; and oral dexamethasone.
  MAINTENANCE THERAPY: Patients receive oral mercaptopurine; oral methotrexate; vincristine IV; and oral dexamethasone.
- MOAD+Campath-Step 2: Campath 10 mg dose
  INDUCTION THERAPY: Patients receive methotrexate IV; vincristine IV and asparaginase IM; oral dexamethasone; and alemtuzumab SC.
  CONSOLIDATION THERAPY: Patients receive methotrexate IV and asparaginase IM.
  CYTOREDUCTION THERAPY: Patients receive vincristine IV and oral methotrexate IV; leucovorin calcium IV; and oral dexamethasone.
  MAINTENANCE THERAPY: Patients receive oral mercaptopurine; oral methotrexate; vincristine IV; and oral dexamethasone.
Arm/Group | MOAD+Campath-Step 1 | MOAD+Campath-Step 2
Serious Adverse Events (participants affected / at risk) | 7/7 | 5/5
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOAD+Campath-Step 1 (N=7) | MOAD+Campath-Step 2 (N=5)
CD4 decreased (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 3
Leukocytes decreased (Investigations) | 7 | 5
Lymphopenia (Investigations) | 5 | 1
Neutrophils decreased (Investigations) | 7 | 4
Platelets decreased (Investigations) | 6 | 4
Atrial tachycardia/PAT (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Weight loss (Investigations) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Abdomen, hemorrhage NOS (Gastrointestinal disorders) | 1 | 0
Respiratory tract hemorrhage NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Infection w/ gr3-4 neut, catheter relate (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, colon (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, lung (Infections and infestations) | 2 | 2
Infection w/ gr3-4 neut, oral cavity (Infections and infestations) | 2 | 0
Infection Gr0-2 neut, heart (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, skin (Infections and infestations) | 1 | 0
Opportunistic infection lymphopenia>=gr1 (Infections and infestations) | 0 | 1
Infection w/ gr3-4 neut, blood (Infections and infestations) | 2 | 2
Infection-other (Infections and infestations) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Ataxia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Neuropathy-motor (Nervous system disorders) | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vision-blurred (Eye disorders) | 1 | 0
Anus, pain (Gastrointestinal disorders) | 1 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Head/headache (Nervous system disorders) | 1 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Oral cavity, pain (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MOAD+Campath-Step 1 (N=7) | MOAD+Campath-Step 2 (N=5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 2
Leukocytes decreased (Investigations) | 3 | 1
Lymphopenia (Investigations) | 2 | 0
Neutrophils decreased (Investigations) | 4 | 0
Platelets decreased (Investigations) | 4 | 0
Hematologic-other (Blood and lymphatic system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Fatigue (General disorders) | 7 | 3
Fever w/o neutropenia (General disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 0
Rigors/chills (General disorders) | 2 | 0
Sweating (Skin and subcutaneous tissue disorders) | 3 | 0
Weight loss (Investigations) | 1 | 0
Fibrinogen decreased (Investigations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0
Injection site reaction (General disorders) | 3 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin-other (Skin and subcutaneous tissue disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Teeth (Gastrointestinal disorders) | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 3 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 3 | 2
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 1
Taste disturbance (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
GI-other (Gastrointestinal disorders) | 1 | 0
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0
Infection w/ gr3-4 neut, oral cavity (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, upper airway (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 2 | 0
Infection Gr0-2 neut, sinus (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, skin (Infections and infestations) | 1 | 0
Edema limb (General disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 6 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Creatinine increased (Investigations) | 3 | 0
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic/Laboratory-other (Investigations) | 3 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 2 | 2
Vision-blurred (Eye disorders) | 2 | 1
Tearing (Eye disorders) | 1 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Head/headache (Nervous system disorders) | 2 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Oral cavity, pain (Gastrointestinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Syndromes-other (General disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less